CLINICAL TRIAL: NCT05922241
Title: Comparative Effects of Costophrenic Assisted Cough and Anterior Chest Compression Technique on Sputum Diary, Oxygen Saturation, Expiratory Flow Rate, and Dyspnea in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Comparative Effects of Costophrenic Assisted Cough and Anterior Chest Compression Technique in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0317
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Anterior chest compression; Chest Physio; Costophrenic assist; Sputum expectoration; Oxygen Saturation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costophrenic assisted cough (Experimental): While doing Costophrenic assist: at the end of expiration, the therapist gives a quick stretch to the diaphragm and intercostals to facilitate more complete inhalation by compressing the chest at the costophrenic angle toward the central tendon of the diaphragm. This is done several times to fill the lungs. The patient is then instructed to hold the air in the lungs. As the patient gets ready to cough, the therapist performs a diaphragmatic assist by applying a strong pressure up and in toward the central tendon
  Interventions: Other: Costophrenic assisted cough
- Anterior chest compression (Experimental): Anterior chest compression: the therapist places one arm across the patient's pectorals and the other parallel to it on the lower abdomen. After the patient takes a maximal breath, the therapist pushes down to help the patient cough. The greatest force is applied through the lower chest during expulsion
  Interventions: Other: Anterior chest compression

INTERVENTIONS:
Other: Costophrenic assisted cough — Therapist places the hands on the costophrenic angles of the patient's rib cage. During the patient's inspiration, the therapist applies a series of three repeated quick-stretch contractions down and in to encourage maximal inspiration. At the end of expiration, the therapist applies a quick stretch down and in on the patient's lower chest to facilitate a stronger diaphragmatic and intercostal muscle contraction. While instructing the patient to cough, the therapist applies strong pressure through the hands in toward the central tendon of the patient's diaphragm
  Arms: Costophrenic assisted cough
Other: Anterior chest compression — The therapist puts one arm across the patient's pectoral region to stabilize or compress the upper chest while the other arm is placed either parallel on the lower chest or abdomen below the xiphoid process
  Arms: Anterior chest compression

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory lung disease that causes obstructed airflow from the lungs. Symptoms include breathing difficulty, cough, mucus (sputum) production and wheezing. In Costophrenic assist, the therapist gives a quick stretch to the diaphragm and intercostals with repetitions. The patientt holds air in the lungs. As the patient gets ready to cough, the therapist performs a diaphragmatic assist. In Anterior chest compression: the therapist places one arm across the patient's pectorals and the other parallel to it. After the patient takes a maximal breath, the therapist pushes down to help the patient cough. The greatest force is applied through the lower chest during expulsion. A total 34 patients will be taken. 2 groups will be created to apply intervention. After signing consent form, 17 patients in group A will be given costophrenic assist technique and 17 patients in group B will be given anterior chest compression technique. Baseline treatment given to both groups will include percussion and tapping. The data collected will then be analyzed using IBM SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

* Stable Patients
* Mild to Moderate Patients of COPD according to gold criteria
* Decreased O2 Saturation Levels
* Immobilized Mucus

Exclusion Criteria:

* Tachycardia
* Tachypnea
* Non Covid
* Cardiovascular Pathology
* Myopathy
* Neurogenic Disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Breathlessness, Cough and Sputum Scale (BCSS) | fourth week
  The breathlessness, cough and sputum scale (BCSS) are a three-item scale that rates symptoms of dyspnea, cough and sputum on a Likert scale from 0 (no symptoms) to 4 (severe symptoms)
Modified Borg Dyspnea (RPE) scale | fourth week
  The most popular tool for evaluating symptoms of breathlessness is the Modified Borg Dyspnoea Scale. RPE scales, despite being a subjective gauge of exercise intensity, are useful when utilised properly. The RPE scale has a 0 to10 scale with 0 being no exertion and 10 being maximum effort
Peak Flow Meter | fourth week
  A peak flow meter must be used by blowing forcefully into it. In liters per minute, the meter measures the forced air flow. When you exhale, the indicator on the device moves and gives you a reading on a scale of 1 to 10. When a person's airway function changes, it may be a sign that their asthma or COPD symptoms are getting worse. This is where a peak flow meter is useful
Pulse Oximeter: | fourth week
  The oxygen saturation level of your blood can be measured with a non-invasive procedure called pulse oximetry. It can quickly identify even minute variations in oxygen levels. These levels demonstrate how well blood transports oxygen to your arms and legs, which are the extremities that are farthest from your heart

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petty TL. The history of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):3-14. doi: 10.2147/copd.2006.1.1.3. PMID 18046898
- [Background] Lopez-Campos JL, Calero C, Quintana-Gallego E. Symptom variability in COPD: a narrative review. Int J Chron Obstruct Pulmon Dis. 2013;8:231-8. doi: 10.2147/COPD.S42866. Epub 2013 May 7. PMID 23687444
- [Background] Arık S, Çevik K. Effect of Postural Drainage and Deep Breathing-Cough Exercises on Oxygen Saturation, Triflo Volume and Pulmonary Function Test in Patients with COPD. Journal of Clinical & Experimental Investigations. 2021;12(4).
- [Background] Ramos FL, Krahnke JS, Kim V. Clinical issues of mucus accumulation in COPD. Int J Chron Obstruct Pulmon Dis. 2014 Jan 24;9:139-50. doi: 10.2147/COPD.S38938. eCollection 2014. PMID 24493923